CLINICAL TRIAL: NCT02136667
Title: Preeclampsia and Circulating Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other); Karen Elise Jensen Foundation (Other); Central Denmark Region (Other)
Responsible Party: Sponsor
Other Study IDs: 98372017
Record Dates: First submitted 2014-05-01; First posted 2014-05-13 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-05

CONDITIONS: Postpartum CVD Risk in Women With Previous Preeclampsia.
Keywords: Preeclampsia; Cardiovascular disease (CVD) risk
MeSH Terms: conditions — Pre-Eclampsia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood serum Blood plasma Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed: Women with a history of preeclampsia 10 years ago
- Unexposed: Women with a history of uncomplicated pregnancy 10 years ago

SUMMARY:
In order to assess circulating biomarkers of cardiovascular risk, we will conduct a 10-year follow-up study comparing 32 exposed (women with a history of pregnancy complicated by preeclampsia) and 32 unexposed (women with a history of uncomplicated pregnancy).

Participants will be recruited from a well-characterised cohort, previously assembled during their pregnancies, at the Department of Obstetrics at Randers Regional Hospital in 2001-2004.

Blood and urine samples, collected during their pregnancies, are stored in a biobank, thus rendering the possibility of longitudinal assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participation in previous study 2001-2005.

Exclusion Criteria:

* Current pregnancy or breastfeeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from a well-characterised cohort, previously assembled at the Department of Obstetrics at Randers Regional Hospital in 2001-2005.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Circulating biomarkers of cardiovascular disease 10 years postpartum. | 10 years postpartum

SECONDARY OUTCOMES:
Markers of arteriosclerosis and atherosclerosis | 10 years postpartum
Circulating biomarkers of cardiovascular disease at baseline pregnancy. | During pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ulla B Knudsen, Professor, Study Chair — Department of Obstetrics and Gynaecology, Aarhus University Hospital; Martin Christensen, MD, Principal Investigator — Clinical Research Unit, Randers Regional Hospital; Camilla S Kronborg, MD, PhD, Study Director — Department of Oncology, Aarhus University Hospital
Locations (1):
- Randers Regional Hospital, Randers, Randers NØ, Denmark